CLINICAL TRIAL: NCT03323489
Title: Celiac Plexus Radio-Surgery for Pain Management in Advanced Cancer Patients - a Phase II Trial
Brief Title: Celiac Plexus Radio-Surgery for Pain Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Yaacov Lawrence (Other Government)
Responsible Party: Sponsor-Investigator, Dr. Yaacov Lawrence, Vice Chair, and Director, Center for Translational Research in Radiation Oncology Dep. Radiation Oncology, Sheba Medical Center
Organization: Sheba Medical Center (Other Government)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHEBA-17-4292-YL-CTIL
Record Dates: First submitted 2017-10-03; First posted 2017-10-27 (Actual); Last update posted 2022-05-12 (Actual); Status verified 2022-05

CONDITIONS: Advanced Cancer; Pancreas Cancer; Pain
Keywords: celiac; radiosurgery; sbrt; radiotherapy; pain
MeSH Terms: conditions — Pancreatic Neoplasms; Pain; Celiac Disease

STUDY DESIGN:
Intervention Model Description: all of the patients will be treated.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- celiac radiosurgery, single fraction (Experimental): Celiac Plexus Radiosurgery
  Interventions: Radiation: Celiac Plexus Radiosurgery

INTERVENTIONS:
Radiation: Celiac Plexus Radiosurgery — patients will receive a single radiation treatment of 25 Gy directed towards the celiac surgery, and at the physician's discretion also abutting tumor

SUMMARY:
Many cancer patients, especially those with pancreatic cancer, suffer from severe lower back / upper abdominal pain. This pain is often poorly managed with standard treatments; the doses of painkiller required often induce side effects, whereas nerve block procedures (where a needle is deeply inserted into the back) are both invasive and of limited benefit.

This clinical trial investigates a unique novel approach in which high-dose radiation (radiosurgery) is focused on the offending nerve bundle (the celiac plexus) in the posterior abdomen. Preliminary results from a single institution pilot trial are very promising: pain relief is substantial and side effects minimal. In this multi-center clinical trial, patients will be accrued and receive treatment at several international locations.

Main aim of the study:

Establish the safety and efficacy of the treatment in the multi-center setting.

This trial will bring pain relief to cancer sufferers and improve current acceptable standard of care. The trial resonates with the Gateway mission of promoting new treatments that directly benefit people living with cancer, enhancing their wellbeing, and consequently decreasing the fear associated with a cancer diagnosis.

DETAILED DESCRIPTION:
Severe lower back pain radiating anteriorly in a belt-like distribution is characteristic of pancreatic cancer. The pain is thought related to involvement of the celiac nerve plexus, located behind the pancreas; due to either macroscopic compression or microscopic perineural invasion.

Contemporary approaches (narcotic analgesics, celiac nerve blocks and systemic chemotherapy) each have drawbacks, and as a consequence many patients suffer from severe pain. We hypothesized that ablative radiosurgery (high dose, precise X-ray treatment) focused on the celiac plexus would succeed in palliating these patients, possibly by interrupting pain transmission. It is important to emphasize that bringing pain relief to cancer patients is not only humane, but also associated with improved mood, quality of life and possibly improved survival. Our preliminary results suggest that the treatment is both effective and well tolerated; furthermore it appears that the patients tolerate subsequent cytotoxic treatments better. We will perform a prospective phase II multicenter clinical trial to test our hypothesis Compared to the small pilot trial the follow-up trial will: 1) Enroll a larger number of patients (n=100). 2) Be performed across a number of institutions, in both the Middle East and the United States. 3) Include improved measures of quality of life and functional capacity. 'Caregiver burden' and 'Patient hope' will also be assessed. 4) Incorporate exploratory translational endpoints relating to immune activation.

Target population Adult patients with severe, poorly controlled lower back/abdominal pain (intensity at least 5/10 on the Numeric Pain Rating Scale) thought to originate in the celiac plexus (generally, but not exclusively, from pancreatic cancer). Patients with a poor prognosis, and those with previous radiation to the upper abdomen will be excluded. Systemic therapies will need to be stopped several days prior to, and following, treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years.
2. ECOG performance status ≤2 (Karnofsky ≥60%, see Appendix A section 24).
3. Patients must have a malignancy that is metastatic or unresectable (for surgical or medical reasons).
4. Typical retroperitoneal pain syndrome (pain that radiates from the lower back to the upper abdomen, belt like distribution).
5. Uncontrolled pain at recruitment, defined as >=5 on 11 point BPI scale despite analgesic use.
6. Anatomical involvement of the celiac plexus, as defined by at least one of the following:

   1. Any Pancreatic cancer
   2. Any other cancer that on imaging demonstrates either: gross involvement of the celiac blood vessels or celiac plexus on imaging OR haziness around the celiac blood vessels, that typically implies tumor engulfment.
7. Recent abdominal imaging (CT, PET or MRI) should be at most 2 months old. The CT simulation performed as part of the protocol will be considered sufficient.
8. Prior chemotherapy or biological treatment is allowed, but any active oncological treatment should be stopped at least 6 days prior to radiation and renewed at least 6 days following radiation. For trastuzumab emtansine a 14 break prior to, and a 6 day break post-therapy is required. Hormonal treatments (e.g. tamoxifen, androgen ablation, androgen antagonists, aromatase inhibitors), and bone-strengthening agents (e.g. bisphosphonates, anti-RANKL antibody denosumab) may be continued during the radiation treatment, and do not need to be interrupted.
9. Willingness to attend 3- and 6- week follow-up visits, and participate in telephone follow-up thereafter.
10. Radiation is known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of therapy.
11. Ability to understand and the willingness to sign a written informed consent document.
12. Before patient registration, written informed consent must be provided.

Exclusion Criteria:

1. Patients under 18 years of age
2. Patients who are well balanced in terms of pain control
3. Patients with life expectancy <8 weeks as defined by the primary oncologist.
4. Known serum albumin <2.4 (does not need to be especially tested if unknown).*
5. Known lymphopenia defined as <12% of white blood count (does not need to be especially tested if unknown).*
6. Altered mental status (defined as change in brain function from baseline including confusion, drowsiness, delirium, dementia or coma)*
7. Leptomeningeal spread*
8. Current or previous spinal cord compression*
9. Significant comorbidities (this is left to physicians' discretion. Guidance provided below section 8.4. As an example, patients with metastatic cancer, in the context of combined impaired renal and hepatic function are expected to have a poor survival)*
10. Patients with ECOG Performance status 3 or 4*
11. Any concurrent chemotherapy or biologic treatment is prohibited during 1 week before until 1 week following radiotherapy.
12. Previous radiotherapy to upper abdomen.
13. Conditions associated with increased side effects to radiotherapy (Inflammatory bowel disease, scleroderma for example).
14. Patients who have not recovered from the acute adverse events due to prior anti-cancer therapy (however peripheral neuropathy and other chronic side effects of anti-cancer therapy are not exclusion criteria).
15. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
16. Special populations: pregnant women, prisoners, patients with major psychiatric illnesses.
17. Unwilling or unable to attend 3-week and 6-week post treatment assessments.

    * these factors are all associated with a very poor prognosis. 40 ------ Nb There are criteria that exclude patients from performing the six-minute walk test (see section 29). These patients may nonetheless participate in the protocol and undergo celiac axis radiosurgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2022-01-30 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Change in Pain level from baseline - as measured using BPI | three weeks
  complete or partial pain response as assessed with the BPI scale

SECONDARY OUTCOMES:
Average Pain Level | 3 weeks and 6 weeks
  Patient reported average pain as assessed with the BPI scale (0 to 10)
Opioid use | 3 weeks and 6 weeks
  daily opioid usage
Quality of Life as measured using FACT-Hep questionnaire | 3 weeks and 6 weeks
  as measured using FACT-Hep scale
six minute walk | 3 weeks and 6 weeks
  assess how far patient can walk in 6 minutes, a measure of functionality
hand grip strength | 3 weeks and 6 weeks
  measure with hand dynamometer, a measure of functionality

CONTACTS AND LOCATIONS:
Locations (7):
- United States (2):
  - The Mount Sinai Hospital, New York, New York
  - The Ohio State University Comprehensive Cancer Center, Columbus, Ohio
- Princess Maragret Cancer Center, Toronto, Ontario, Canada
- Israel (3):
  - Sheba Medical Center, Ramat Gan
  - Assuta Hospital in Ramat HaHayal, Tel Aviv
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Instituto Português de Oncologia do Porto Francisco Gentil, Porto, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lawrence YR, Miszczyk M, Dawson LA, Diaz Pardo DA, Aguiar A, Limon D, Pfeffer RM, Buckstein M, Barry AS, Meron T, Dicker AP, Wydmanski J, Zimmermann C, Margalit O, Hausner D, Morag O, Golan T, Jacobson G, Dubinski S, Stanescu T, Fluss R, Freedman LS, Ben-Ayun M, Symon Z. Celiac plexus radiosurgery for pain management in advanced cancer: a multicentre, single-arm, phase 2 trial. Lancet Oncol. 2024 Aug;25(8):1070-1079. doi: 10.1016/S1470-2045(24)00223-7. Epub 2024 Jul 16. PMID 39029483
- [Derived] Jacobson G, Fluss R, Dany-BenShushan A, Golan T, Meron T, Zimmermann C, Dawson LA, Barry A, Miszczyk M, Buckstein M, Diaz Pardo D, Aguiar A, Hammer L, Dicker AP, Ben-Ailan M, Morag O, Hausner D, Symon Z, Lawrence YR. Coeliac plexus radiosurgery for pain management in patients with advanced cancer : study protocol for a phase II clinical trial. BMJ Open. 2022 Mar 24;12(3):e050169. doi: 10.1136/bmjopen-2021-050169. PMID 35332036